CLINICAL TRIAL: NCT05239273
Title: Investigation of the Effects of Complex Decongestive Therapy Applied on Patients With Lower Extremity Lymphedema on Body Awareness, Functionality and Quality of Life
Brief Title: Effects of Complex Decongestive Therapy Applied on Patients With Lower Extremity Lymphedema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, seyda toprak celenay, associate professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/02/05
Record Dates: First submitted 2022-02-05; First posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complex Decongestive Therapy (CDT) Group (Experimental): Phase 1 of CDT will be applied to CDT group. This application consists of manual lymph drainage, skin care, compression bandage and exercises. This phase will continue 5 days a week for 3 weeks.
  Interventions: Other: Complex Decongestive Therapy
- Control group (Other): Waiting list will included in control group.
  Interventions: Other: Control

INTERVENTIONS:
Other: Complex Decongestive Therapy — Phase 1 of CDT will be applied. This application consists of manual lymph drainage, skin care, compression bandage and exercises.
  Arms: Complex Decongestive Therapy (CDT) Group
Other: Control — No intervention
  Arms: Control group

SUMMARY:
The aim of this study is to investigate the effects of complex decongestive therapy applied to patients with lymphedema in the lower extremities on body awareness, functionality and quality of life.

DETAILED DESCRIPTION:
Lymphedema is a chronic condition characterized by the permanent accumulation of protein-rich fluid in certain body regions as a result of the dysfunction of the lymphatic system, in which skin and subcutaneous changes are added to the picture. Pain in the affected extremity and other accompanying lymphedema symptoms can negatively affect functionality and quality of life, and swelling in the extremity can negatively affect the body image of individuals. Today, Complex Decongestive Therapy (CDT) is accepted as the gold standard in the treatment of lymphedema. It has been shown in the literature that CDT has positive effects on parameters such as functionality, quality of life, and balance in patients with upper limb lymphedema. There are few studies investigating the effects of CDT on body awareness, functionality and quality of life in patients who developed lymphedema in the lower extremities.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-65
* Having unilateral lymphedema in the lower extremity
* Volunteer to participate in the study

Exclusion Criteria:

* Having bilateral lower extremity lymphedema
* Having an active infection
* Having a mental cognitive disorder
* Being unable to communicate and cooperate
* Conditions where manual lymphatic drainage is contraindicated (such as severe heart failure and/or uncontrolled rhythm disturbance, uncontrollable hypertension, being pregnant, presence of thrombus, active infection ect.)
* Presence of metastases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Body Awareness | change from baseline at 3 weeks
  Body Awareness Questionnaire will be used to assess body awareness. This questionnaire was developed by Mallory & Simon and has Turkish validity and reliability. The survey consists of 18 questions. The total score ranges from 18 to 126. As the total score increases, it is concluded that body awareness is good.

SECONDARY OUTCOMES:
Lower Extremity Functionality | change from baseline at 3 weeks
  Lower extremity functionality will be evaluated with the Lower Extremity Functional Scale. The lower extremity functional scale consists of 20 items and each item is scored between 0-4 and evaluated in 5 items. These are frequently: extreme difficulty/inability to perform the activity, quite difficult, moderate difficulty, a little difficulty and no difficulty. The total score ranges from 0 to 80, and higher scores represent better functional level
Life quality | change from baseline at 3 weeks
  Life quality will be assessed by the Lymphedema Quality of Life Questionnaire. The questionnaire, which consists of 21 questions, consists of the subheadings of Function, Body Image, Symptom, and Emotion. It has a score ranging from 1 to 4 for the first 20 questions. The total score for each area is calculated by adding all the scores and dividing by the total number of questions answered. High scores indicate lower quality of life. The last question about general quality of life is scored between 0 and 10.
Edema evaluation | change from baseline at 3 weeks
  Edema evaluation will be made with circumference measurement from the lateral malleolus to the groin at intervals of 4 cm.

CONTACTS AND LOCATIONS:
Overall Officials: Seyda Toprak Celenay, Principal Investigator — Ankara Yildirim Beyazıt University